CLINICAL TRIAL: NCT05472285
Title: Evaluation of the Effects of a Food Supplementation on the Improvement of Cognitive Functions in Healthy Seniors: a Randomized Double-blind Study Versus Placebo
Brief Title: Evaluation of the Effects of a Food Supplementation on the Improvement of Cognitive Functions in Healthy Seniors
Acronym: BioMind
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bionov (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2021-A02122-39
Record Dates: First submitted 2022-07-19; First posted 2022-07-25 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2022-07

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Intervention Model Description: This study is designed as a multicentric, randomized, parallel arms, double-blind, placebo-controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Active Comparator): 2 capsules per day during 8 weeks
  Interventions: Dietary Supplement: Verum
- Placebo (Placebo Comparator): 2 capsules per day during 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Verum — After randomization (visit V1), subjects will consume orally 2 capsules per day, during the breakfast, for 8 weeks (from visit V1 to visit V3).
  Arms: Verum
Dietary Supplement: Placebo — After randomization (visit V1), subjects will consume orally 2 capsules per day, during the breakfast, for 8 weeks (from visit V1 to visit V3).
  Arms: Placebo

SUMMARY:
The hypothesis of this study is to evaluate the effect of supplementation for 8 weeks on the improvement of cognitive functions in healthy seniors with or without mild cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Age between 55 and 70 years (limits included),
* Subjects with mild cognitive decline (MMSE between 21 and 24, including bounds) and healthy (MMSE >24 to 30).
* Subject with a Hamilton Anxiety Scale score between 5 and 17 (limits included),
* BMI between 18.5 and 29.5 kg/m² (limits included),
* Menopausal woman without hormone replacement therapy (at least 12 months without menstruation),
* Stable diet for at least 3 months,
* Blood pressure below 14/90 mm HG,
* With no significant change in dietary habits or physical activity during the 3 months preceding randomization and agreeing to maintain them unchanged throughout the study,
* Good general and mental health with in the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or physical examination,
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form,
* Affiliated with a social security scheme,
* Agree to be registered on the volunteers in biomedical research file.

Exclusion Criteria:

* Suffering from a metabolic disorder such as diabetes treated or not, uncontrolled thyroidal trouble or other metabolic disorder,
* Suffering from a serious chronic disease (cancer (ongoing and if in remission for less than 5 years), HIV, renal failure, ongoing biliary or liver disorder, psychiatric pathologies (bi-polar disorders, depression, degenerative brain diseases (Alzheimer, vascular dementia, etc.), immunodeficiency, uncontrolled heart disease, arthritis, chronic respiratory disorder, chronic inflammatory digestive disease or a gastrointestinal disorder deemed incompatible with driving the vehicle. ), immunodeficiency, uncontrolled heart disease, arthritis, chronic respiratory disorder, chronic inflammatory digestive disease or a gastrointestinal disorder deemed incompatible with the conduct of the study by the investigator (e.g. celiac disease, Crohn's disease, irritable bowel disease, etc.).
* For Women: Non-menopausal woman or menopausal woman with hormone replacement therapy
* Consuming more than 5 cigarettes per day,
* With a known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredient,
* Under antioxidant treatment (vitamin A, C, E, β-carotene, lutein, lycopene, selenium, Ginkgo biloba, dehydroepiandrosterone, polyphenol in the broad sense, phytoestrogen, ...), sedative drugs (neuroleptics, benzodiazepines, anxiolytics, hypnotics) and related drugs, antidepressants, antipsychotics, mood stabilizers, (hypnotic anti-histamines... ), cognitive treatment or dietary supplements that could affect the parameters monitored during the study in the opinion of the investigator or in the month preceding the V1 visit.
* Volunteer consuming no more than 400mg/d of total caffeine in a day (addition of beverages such as coffee, tea, energy drinks and soft drinks), [6 espressos = 162mg of caffeine and 4 mugs of filter coffee = 380mg, 8 cups of black tea = 360mg].
* Having a consumption of herbal infusions or waters > 2 liters / day
* Presenting a high probability of non-compliance with the protocol or of dropping out during the study (geographical instability, insufficient motivation, psychological profile, etc),
* Drinking more than 2 glasses of alcohol per day, every day and without interruption, and not willing to keep their drinking habits unchanged throughout the study
* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial
* Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros,
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision,
* Presenting a psychological or linguistic incapability to sign the informed consent,
* Impossible to contact in case of emergency.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
The change in mental fatigue | up to 10 weeks
  Mental fatigue is assessed twice on a VAS (Visual Analogue Scale) in the COMPASS test, which is a computerized test assessing cognitive functions. The first VAS is assessed following the cognitive Demand Battery comprising 3 tasks, namely a 3s serial subtraction task, a 7s serial subtraction task and another COMPASS task called Digit vigilance.

SECONDARY OUTCOMES:
Evolution of global cognitive functioning | up to 10 weeks
  Assessed with MMSE score
Evolution of cognitive function | up to 10 weeks
  Assessed with COMPASS score
The frequency of adverse events | up to 10 weeks
  The frequency of subjects with at least one AE (Adverse Event), SAE (Serious Adverse Event), treatment-emergent AE and treatment-emergent SAE and the number of corresponding events

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinical Investigation Unit Biofortis - Paris, Paris
  - Clinical Investigation Unit of Biofortis - SHE, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No